CLINICAL TRIAL: NCT01990911
Title: Renal Sympathetic Denervation Restores Autonomic Imbalance and Prevents Atrial Fibrillation in Patients With Hypertensive Heart Disease: a Pilot Study
Brief Title: Renal Sympathetic Denervation Prevents Atrial Fibrillation in Patients With Hypertensive Heart Disease: a Pilot Study
Acronym: RDPAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pace Clinic (Other)
Collaborators: University Hospital, Saarland (Other)
Responsible Party: Principal Investigator, Marshall Jacobus Heradien, Dr, Pace Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RDPAF1
Record Dates: First submitted 2013-11-09; First posted 2013-11-25 (Estimated); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Hypertension; Hypertensive Heart Disease; Atrial Fibrillation; Autonomic Imbalance
Keywords: hypertension; hypertensive heart disease; atrial fibrillation; autonomic imbalance
MeSH Terms: conditions — Hypertension; Atrial Fibrillation | interventions — Nutrition Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal denervation (Experimental): Renal denervation: both renal arteries are denervated by applying radio-frequency energy at application points moving in a helical fashion starting in the distal renal artery and moving to the proximal junction with the abdominal aorta.
  Interventions: Device: Renal denervation; Drug: Medical therapy
- Medical therapy (Sham Comparator): This group will not receive renal sympathetic denervation
  Interventions: Drug: Medical therapy

INTERVENTIONS:
Device: Renal denervation — In patients randomized to intervention both renal arteries will be treated with radio-frequency energy as per standard Symplicity protocol.In patients randomized to medical-treatment group only, sham renal denervation will be performed by only injecting contrast agent into both renal arteries.
  Other Names: Symplicity catheter renal denervation
  Arms: Renal denervation
Drug: Medical therapy — Subjects will continue on their standard medical therapy as prescribed by their treating physician
  Other Names: Three or more blood pressure tablets, including a diuretic

SUMMARY:
The autonomic nervous system plays an important role in the precipitation of AF in structurally-abnormal hearts. Restoration of autonomic imbalance may therefore prevent new-onset AF.

Renal artery denervation (RDN) is a novel percutaneous procedure that uses radio-frequency energy to destroy the sympathetic renal nerves. Symplicity 1 and -2 studies have shown that RDN effectively reduces blood pressure in up to 80% of treated patients. LVH regression and improvement of diastolic dysfunction follow as a consequence of afterload reduction and renin-angiotensin-aldosterone system modulation. RDN may thus also reduce intra-atrial pressure resulting in less stretch of the pulmonary venous ostia where most ectopic AF-foci originate.

Hypothesis: RDN restores autonomic imbalance in HTHD and lowers intra-atrial pressure by reducing afterload. These synergistic mechanisms may prevent new-onset AF.

DETAILED DESCRIPTION:
One hundred consenting patients meeting all inclusion criteria will undergo an exercise stress test, 2D and M-Mode echocardiograms and 24-hour ambulatory blood pressure holter monitoring prior to being randomised to receive either renal denervation (RDN) with a Symplicity renal denervation catheter plus medical therapy or medical therapy alone. Coronary angiography with/without coronary revascularisation will be performed as per the treating cardiologist's clinical judgement and a Reveal® holter will be implanted in all patients at the end of the procedure.

Time zero will be defined as starting at three months after the procedure. Follow up visits will be scheduled to scan the holter for the primary end point, i.e. high atrial rates (AF-surrogate defined as: "episodes of atrial rate >190 beats per minute for more than 6 minutes") or new-onset AF. Patients will be followed six monthly for three years.

ELIGIBILITY:
Inclusion Criteria:

* Must have an indication for coronary angiography e.g.
* Acute coronary syndrome
* Positive stress ECG: - Defined as ≥1mm ST segment shift (depression or elevation) in ≥2 contiguous leads with/without chest discomfort)
* Age ≥55 years
* Office blood pressure ≥160/90mmHg in non-diabetics or ≥150/90mmHg in diabetics
* Subjects must be on at least 3 anti-hypertensive drugs, including a diuretic agent
* Sinus rhythm
* Left ventricular hypertrophy defined on echo as:
* Estimated LV mass > 255 g or LVMI >131 g/m2 for men
* Estimated LV mass >193 g or LVMI >113 g/m2for women
* Left atrial diameter ≥45mm on any echocardiographic window

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) < 45ml/min/1.73m2
* Renal artery anatomy unsuitable for RDN
* Substantial stenotic valvular heart disease
* Pregnancy or planned pregnancy
* Thyrotoxicosis
* Patients needing to undergo coronary artery bypass surgery

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation | 3 years
  Subclinical atrial tachyarrhythmias (episodes of atrial rate >190 beats per minute for more than 6 minutes) or atrial fibrillation recorded by implantable loop recorder (Reveal® holter).

SECONDARY OUTCOMES:
Restoration of autonomic imbalance | 3 years
  Restoration of autonomic imbalance: lowering resting heart rate, prolonging the PR-interval and improving heart rate recovery after exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Brink, PhD, Study Director — Tygerberg Hospital and Stellenbosch University; Michael Bohm, PhD, Study Director — University Hospital, Saarland
Locations (1):
- Pace Clinic, Cape Town, Western Cape, South Africa

REFERENCES:
- [Background] Heradien M, Mahfoud F, Greyling C, Lauder L, van der Bijl P, Hettrick DA, Stilwaney W, Sibeko S, Jansen van Rensburg R, Peterson D, Khwinani B, Goosen A, Saaiman JA, Ukena C, Bohm M, Brink PA. Renal denervation prevents subclinical atrial fibrillation in patients with hypertensive heart disease: Randomized, sham-controlled trial. Heart Rhythm. 2022 Nov;19(11):1765-1773. doi: 10.1016/j.hrthm.2022.06.031. Epub 2022 Jun 30. PMID 35781044